CLINICAL TRIAL: NCT00233662
Title: An Open-Label, Multicenter Study to Evaluate the Safety and Tolerability of Repeat Courses of Intramuscular Administration of Alefacept (LFA-3/IgG1 Fusion Protein) in Patients With Chronic Plaque Psoriasis
Brief Title: Safety and Tolerability of Repeat Courses of IM Alefacept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-733
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Alefacept

INTERVENTIONS:
Drug: Alefacept

SUMMARY:
The purpose of this study is to determine whether repeat courses of alefacept, administered intramuscularly, are safe when given to chronic plaque psoriasis patients who are receiving standard dermatology treatments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* At least 16 years of age.
* Diagnosed with chronic plaque psoriasis and require systemic therapy.
* CD4+ lymphocyte counts at or above the lower limit of normal for Covance Central Laboratory Services, Inc., unless on a stable dose of prednisone (counts must be at or above 300 cells/mm3).

Exclusion Criteria:

* Unstable erthrodermic or pustular psoriasis.
* Diagnosis of guttate psoriasis.
* Serious local infection or systemic infection within 3 months prior to first dose of alefacept.
* Positive for HIV antibody.
* Known invasive malignancy within 5 years of enrollment. Patients with a history of treated squamous cell and/or basal cell carcinomas limited to the skin are not excluded.
* Evidence of active tuberculosis.
* Current treatment for active tuberculosis or tuberculosis prophylaxis.
* Female patients unwilling to practice effective contraception as defined by the investigator.
* Female patients who are pregnant or breast-feeding.
* Current enrollment in any other investigational drug study.
* Previous participation in this study or previous alefacept studies.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2002-12-01 (Actual); Study Completion 2005-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of infections, malignancies, serious adverse events, adverse events leading to discontinuation of study drug, dose withholding (due to infection or decreased T cells), and changes in lymphocyte counts over time.

SECONDARY OUTCOMES:
Patients who achieve a Physician Global Assessment (PGA) of "almost clear" or "clear" over time; the duration of the response to alefacept (the amount of time after alefacept treament before re-treatment with alefacept is necessary).

CONTACTS AND LOCATIONS:
Overall Officials: Barry Ticho, MD, Study Director — Biogen; Kenneth Gordon, MD, Principal Investigator — Loyola University
Locations (46):
- United States (19):
  - University of California, Irvine, Irvine, California
  - University of California, San Francisco, San Francisco, California
  - Clinical Research Specialists, Inc., Santa Monica, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Loyola University Medical Center, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Central Dermatology, St Louis, Missouri
  - University of Medicine and Dentistry Robert Wood Jonhson Medical School, New Brunswick, New Jersey
  - New York University School of Medicine, New York, New York
  - The Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Baylor Dermatology Research Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
- University of Vienna, Vienna, Austria
- Canada (5):
  - Western Canada Dermatology Institute, Edmonton, Alberta
  - Vancouver Hospital, Vancouver, British Columbia
  - Eastern Canada Cutaneous Research Associates, Halifax, Nova Scotia
  - Dermatrials Research, Hamilton, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Marselisborg Hospital, Aarhus C, Denmark
- France (4):
  - CHU Henri Mondor, Créteil
  - Hopital L'Archet II, Nice
  - Hospital Saint Louis, Université Paris VII, Paris
  - Hopital Lyon Sud, Pierre-Bénite
- Germany (11):
  - Humboldt Universitätsklinikum Charité, Berlin
  - St. Josef-Hospital, Bochum
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Heinrich-Heine-Universität, Düsseldorf
  - J W Goethe Universität, Frankfurt
  - Klinikum der Albert-Ludwig-Universität, Freiburg im Breisgau
  - Universitäts Kliniken, Göttingen
  - Universitätskrankenhaus Eppendorf, Hamburg
  - Universitätskliniken des Saarlandes, Homburg/Saar
  - Universität Mannhein, Mannheim
  - Universitätsklinikum Münster, Münster
- Netherlands (2):
  - AMC University of Amsterdam, Amsterdam
  - University Hospital Nijmegen - St. Radboud, Nijmegen
- Hospital Cantonal, Geneva, Switzerland
- United Kingdom (2):
  - St. John's Institute of Dermatology, London
  - Academic Dermatology, Salford